CLINICAL TRIAL: NCT05145322
Title: In Vivo Assessment of the Tooth-Resin Composite Interface Using Optical Coherence Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00011286
Record Dates: First submitted 2021-10-12; First posted 2021-12-06 (Actual); Results first posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Cavity; Cavities of Teeth
Keywords: Dental Composite
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group 1 (Experimental): Group 1: Lesion-specific cavity design with 90 degree cavosurface angle throughout the cavity margins
  Interventions: Device: Composite with 90 degree cavosurface angle
- Group 2 (Experimental): Lesion-specific cavity design with wide bevel throughout the cavity margins
  Interventions: Device: Composite with wide bevel

INTERVENTIONS:
Device: Composite with 90 degree cavosurface angle — Lesion-specific cavity design with 90 degree cavosurface angle throughout the cavity margins will be prepared. The total etch method will be performed, i.e. with a 32% by weight phosphoric acid (3M Scotchbond™ Universal Etchant) on enamel and dentine for 15 seconds. The etchant will be rinsed away and an adhesive (3M Scotchbond™ Universal Adhesive) will be applied on dentine with a microbrush for 20 seconds. The adhesive will be light-cured for 10 sec with the Elipar S10 curing light (3M Oral Care). Subsequently the preparation will be restored with a bulkfill resin composite (3M Filtek™ One Bulk Fill Restorative) and cured for 20 seconds.
  Arms: Group 1
Device: Composite with wide bevel — Lesion-specific cavity design with wide bevel throughout the cavity margins will be prepared. The total etch method will be performed, i.e. with a 32% by weight phosphoric acid (3M Scotchbond™ Universal Etchant) on enamel and dentine for 15 seconds. The etchant will be rinsed away and an adhesive (3M Scotchbond™ Universal Adhesive) will be applied on dentine with a microbrush for 20 seconds. The adhesive will be light-cured for 10 sec with the Elipar S10 curing light (3M Oral Care). Subsequently the cavity will be restored in with a pre-warmed (using Bioclear Heatsync Kit) bulkfill resin composite (3M Filtek™ One Bulk Fill Restorative) and cured for 20 seconds.
  Arms: Group 2

SUMMARY:
The aim of the study is to compare the short-term marginal integrity of two preparation techniques for Class I composite restoration using two visual assessment techniques, the FDI World Dental Federation and US Public Health Service assessment criteria. In addition, Optical Coherence Tomography (OCT) will be used to assess the marginal integrity of the restoration.

DETAILED DESCRIPTION:
A recent review on clinical studies published on the performance of posterior composite restorations that were recalled at least up to 24-months reported that the overall failure rates for studies conducted between 2006-2016 was 13.13% and the two main reasons for failure in these two decades remained the same, i.e. secondary caries (25.68% - 29.47%) and composite fracture (28.84% - 39.07%). In in vitro studies, secondary caries has been attributed to interfacial gap or marginal defect both of which are consequences of polymerization contraction stresses. However, to date no clinical study has been able to directly establish a link between these stresses (and its consequences) to secondary caries. World Dental Federation (FDI) and United States Public Health Service (USPHS) clinical assessment criteria are the two main systems used to evaluate dental restorations in clinical trials. Both systems are designed to evaluate different properties of a restoration and properties pertaining to marginal integrity has been reported to be the most frequent properties investigated of a resin composite restoration. The grading descriptions for these properties are subjective and the discrimination between grading and between properties (especially between marginal stains and secondary caries) are problematic. Reasons to the lack of such a link is the discriminative deficiency of the clinical visual evaluation systems, the FDI and USPHS assessment criteria, and the ethical dilemma of restoration removal to assess for presence or absence of secondary caries. It has been long acknowledged that an objective clinical measuring tool and new clinical study designs for secondary caries is needed to further the understanding of secondary caries initiation and progression and how these relates to the marginal integrity of dental restorations. This brings forth the need of a sensitive yet clinically applicable assessment method for interfacial debonding and demineralization. Optical coherence tomography (OCT) is an optical, nondestructive and clinically- applicable technique that uses near infra red-light waves to provide cross-sectional images of structures. It is regarded as a standard-of-care equipment in ophthalmology and its clinical application has recently expanded to cardiology and dermatology. In dentistry, it has been used intra-orally in clinical trials to detect and quantify enamel demineralization and to detect mucosal and submucosal lesions. Optical coherence tomography and has been used to assess the performance of dental adhesives in a 12-month in vivo trial on non-carious cervical lesion. The authors reported that OCT outcome measures detected significant differences between groups while visual assessments did not. Hence supplementing the two visual assessment techniques with OCT outcome measures is expected to increase the sensitivity of short term interfacial debonding and demineralization changes. The aim of the study is to compare the short-term marginal integrity of two preparation techniques for Class I composite restoration using two visual assessment techniques, the FDI World Dental Federation and US Public Health Service assessment criteria. In addition, Optical Coherence Tomography (OCT) will be used to assess the marginal integrity of the restoration.

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Fair oral hygiene
* At least 20 teeth in occlusion
* Available for the duration of the study

Tooth-level inclusion Criteria:

* Participants with occlusal caries lesion/s in permanent posterior dentition except wisdom teeth
* Caries lesion can be primary or secondary caries.
* Caries lesion is in the International Caries Detection and Assessment System (ICDAS) 4 or 5 category.
* The extent of the caries lesion bucco-lingually is likely not to exceed two-thirds of the occlusal table.
* The selected tooth must be able to be isolated with either rubber dam or other isolation technique during clinical procedure.
* The selected tooth must have an opposing antagonist.
* The selected tooth should be periodontally healthy.

Exclusion Criteria:

- Signs of bruxism

Tooth-level exclusion criteria:

* Wisdom teeth
* Present with irreversible pulpitis.
* Periodontally compromised tooth that may require extraction.
* Caries lesions that would require cuspal coverage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hooi Pin Chew, BDS, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation: clinical criteria for the evaluation of direct and indirect restorations-update and clinical examples. Clin Oral Investig. 2010 Aug;14(4):349-66. doi: 10.1007/s00784-010-0432-8. Epub 2010 Jul 14. PMID 20628774
- [Background] Ryge G, Snyder M. Evaluating the clinical quality of restorations. J Am Dent Assoc. 1973 Aug;87(2):369-77. doi: 10.14219/jada.archive.1973.0421. No abstract available. PMID 4515696
- [Background] Nazari A, Sadr A, Shimada Y, Tagami J, Sumi Y. 3D assessment of void and gap formation in flowable resin composites using optical coherence tomography. J Adhes Dent. 2013 Jun;15(3):237-43. doi: 10.3290/j.jad.a28623. PMID 23534012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on referral from the dental clinics of the School of Dentistry University of Minnesota and enquiries from the public upon seeing flyers pasted at the Malcolm Moos Tower. The first and last participant were enrolled on 09/23/2021 and 7/15/22 respectively.
Pre-assignment Details: Upon referral from the dental clinic or enquiries, potential participants were invited to attend a telemeeting where the participants were presented with the information of the trial using a MS Powerpoint slide deck. 46 participants were invited to the telemeeting and also attended an in-person screening session to determine whether they meet the inclusion criteria of the study. 36 met the inclusion criteria and were successfully enrolled into the study.
Groups:
- 90-degree Cavosurface Angle Cavity Margin: Group 1: Lesion-specific cavity design with 90 degree cavosurface angle throughout the cavity margins
  Composite with 90 degree cavosurface angle: Lesion-specific cavity design with 90 degree cavosurface angle throughout the cavity margins will be prepared. The total etch method will be performed, i.e. with a 32% by weight phosphoric acid (3M Scotchbond™ Universal Etchant) on enamel and dentine for 15 seconds. The etchant will be rinsed away and an adhesive (3M Scotchbond™ Universal Adhesive) will be applied on dentine with a microbrush for 20 seconds. The adhesive will be light-cured for 10 sec with the Elipar S10 curing light (3M Oral Care). Subsequently the preparation will be restored with a bulkfill resin composite (3M Filtek™ One Bulk Fill Restorative) and cured for 20 seconds.
- Wide-bevel Cavity Margin: Lesion-specific cavity design with wide bevel throughout the cavity margins
  Composite with wide bevel: Lesion-specific cavity design with wide bevel throughout the cavity margins will be prepared. The total etch method will be performed, i.e. with a 32% by weight phosphoric acid (3M Scotchbond™ Universal Etchant) on enamel and dentine for 15 seconds. The etchant will be rinsed away and an adhesive (3M Scotchbond™ Universal Adhesive) will be applied on dentine with a microbrush for 20 seconds. The adhesive will be light-cured for 10 sec with the Elipar S10 curing light (3M Oral Care). Subsequently the cavity will be restored in with a pre-warmed (using Bioclear Heatsync Kit) bulkfill resin composite (3M Filtek™ One Bulk Fill Restorative) and cured for 20 seconds.
Period: Overall Study
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Started | 18 | 18
Restoration Placement | 18 | 18
6-months Follow up | 16 | 17
Completed (Completion is defined as having attended the 18-months follow-up visit.) | 14 | 13
Not Completed | 4 | 5
Not completed — Lost to Follow-up | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.56 (14.51) | 30.17 (7.85) | 31.36 (11.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 5 | 8 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Marginal Staining: World Dental Federation (FDI) Criteria - Baseline
Description: The World Dental Federation (FDI) criteria is 5-point ordinal scale with a score of 5 indicating the worst marginal staining.
  1. No marginal staining
  2. Minor marginal staining, easily removable by polishing.
  3. Moderate marginal staining, not esthetically unacceptable.
  4. Pronounced marginal staining; major intervention necessary for improvement
  5. Deep marginal staining, not accessible for intervention.
  Outcome will be reported as a single score at baseline.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 18 | 18
Participants
  Score 1 | 18 | 18
  Score 2 | 0 | 0
  Score 3 | 0 | 0
  Score 4 | 0 | 0
  Score 5 | 0 | 0

2. Primary Outcome: Marginal Staining: World Dental Federation (FDI) Criteria - 6 Months Follow-up
Description: The World Dental Federation (FDI) criteria is 5-point ordinal scale with a score of 5 indicating the worst marginal staining.
  1. No marginal staining
  2. Minor marginal staining, easily removable by polishing.
  3. Moderate marginal staining, not esthetically unacceptable.
  4. Pronounced marginal staining; major intervention necessary for improvement
  5. Deep marginal staining, not accessible for intervention.
  Outcome will be reported as a single score at 6 months post-operative.
Time Frame: 6 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 16 | 17
Participants
  Score 1 | 16 | 17
  Score 2 | 0 | 0
  Score 3 | 0 | 0
  Score 4 | 0 | 0
  Score 5 | 0 | 0

3. Primary Outcome: Marginal Staining: World Dental Federation (FDI) Criteria - 18 Months Follow-up
Description: The World Dental Federation (FDI) criteria is 5-point ordinal scale with a score of 5 indicating the worst marginal staining.
  1. No marginal staining
  2. Minor marginal staining, easily removable by polishing.
  3. Moderate marginal staining, not esthetically unacceptable.
  4. Pronounced marginal staining; major intervention necessary for improvement
  5. Deep marginal staining, not accessible for intervention.
  Outcome will be reported as a single score at 18 months post-operative.
Time Frame: 18 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 14 | 13
Participants
  Score 1 | 14 | 13
  Score 2 | 0 | 0
  Score 3 | 0 | 0
  Score 4 | 0 | 0
  Score 5 | 0 | 0

4. Primary Outcome: Marginal Staining: United States Public Health Service (USPHS) Criteria - Baseline
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst staining.
  A) None. B) Superficial staining (removable, usually localized). C) Deep staining (not removable, generalized).
  Outcome will be reported as a single score at baseline.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Participants
  Score A | 18 | 18
  Score B | 0 | 0
  Score C | 0 | 0

5. Primary Outcome: Marginal Staining: United States Public Health Service (USPHS) Criteria - 6 Months Follow-up
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst staining.
  A) None. B) Superficial staining (removable, usually localized). C) Deep staining (not removable, generalized).
  Outcome will be reported as a single score at 6 months post-operative.
Time Frame: 6 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 16 | 17
Participants
  Score A | 16 | 17
  Score B | 0 | 0
  Score C | 0 | 0

6. Primary Outcome: Marginal Staining: United States Public Health Service (USPHS) Criteria - 18 Months Follow-up
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst staining.
  A) None. B) Superficial staining (removable, usually localized). C) Deep staining (not removable, generalized).
  Outcome will be reported as a single score at 18 months post-operative.
Time Frame: 18 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 14 | 13
Participants
  Score A | 14 | 13
  Score B | 0 | 0
  Score C | 0 | 0

7. Primary Outcome: Marginal Defect: World Dental Federation (FDI) Criteria - Baseline
Description: The World Dental Federation (FDI) criteria is 5-point ordinal scale with a score of 5 indicating the worst marginal defect.
  1. Harmonious outline, no gaps.
  2. Slight ditching, slight step/flashes, minor irregularities.
  3. Major irregularities, ditching or flash, steps
  4. Larger irregularities or steps (repair necessary)
  5. Generalized major gaps or irregularities.
  Margins were assessed quantitatively as 2 different proportions (100% and <100%) of the total length of the margin that is of Score 1 quality.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Participants
  100% of Score 1 | 7 | 8
  <100% Score 1 | 11 | 10

8. Primary Outcome: Marginal Defect: World Dental Federation (FDI) Criteria - 6 Months Follow-up
Description: as for outcome 7
Time Frame: 6 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 16 | 17
Participants
  100% Score 1 | 12 | 12
  <100% Score 1 | 4 | 5

9. Primary Outcome: Marginal Defect: World Dental Federation (FDI) Criteria - 18 Months Post-operative
Description: as for outcome 7
Time Frame: 18 months post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 14 | 13
Participants
  100% Score 1 | 8 | 7
  80 - 99 % Score 1 | 6 | 6

10. Primary Outcome: Marginal Defect: United States Public Health Service (USPHS) Criteria - Baseline
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst defect.
  A) Undetectable. B) Detectable - V-shaped defect in enamel only and catches explorer going both ways.
  C) Detectable - V-shaped defect to the dentin-enamel junction
  Outcome will be reported as a single score at baseline.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Participants
  Score A | 18 | 18
  Score B | 0 | 0
  Score C | 0 | 0

11. Primary Outcome: Marginal Defect: United States Public Health Service (USPHS) Criteria - 6 Months Follow-up
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst defect.
  A) Undetectable. B) Detectable - V-shaped defect in enamel only and catches explorer going both ways.
  C) Detectable - V-shaped defect to the dentin-enamel junction
  Outcome will be reported as a single score at 6 months post-operative.
Time Frame: 6 months Follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 16 | 17
Participants
  Score A | 16 | 17
  Score B | 0 | 0
  Score C | 0 | 0

12. Primary Outcome: Marginal Defect: United States Public Health Service (USPHS) Criteria - 18 Months Post-operative
Description: The United States Public Health Service (USPHS) criteria is 3-point ordinal scale with the 'C' indicating the worst defect.
  A) Undetectable. B) Detectable - V-shaped defect in enamel only and catches explorer going both ways.
  C) Detectable - V-shaped defect to the dentin-enamel junction
  Outcome will be reported as a single score at 18 months post-operative.
Time Frame: 18 months post-operative
Measure: Count of Participants; unit: Participants
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 14 | 13
Participants
  Score A | 14 | 13
  Score B | 0 | 0
  Score C | 0 | 0

13. Secondary Outcome: Backscattered Intensity at the Occlusal Cavosurface Angle.
Description: Presence of elevated intensity at the cavosurface angle (margins) of the restoration, which indicates presence of minor marginal defect, is computed as percentage area of the outline of restoration at every evaluation time point, i.e. baseline, 6 months and 18 months post-operative. Outcome is reported in units of percentage area.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Percentage area
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Percentage area | 6.75 (6.36) | 1.56 (4.33)

14. Secondary Outcome: Tooth-resin Interface Gap at the Occlusal Cavosurface Angle.
Description: Presence of tooth-resin interface gap of more than 0.1 mm at the cavosurface angle (margins) of the restoration, which indicates presence of moderate marginal defect, will be computed as percentage area of the outline of restoration at every evaluation time point, i.e. baseline, 6 months and 18 months post-operative. Outcome is reported in units of percentage area.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Percentage | 14.44 (4.36) | 18.75 (17.63)

15. Secondary Outcome: Backscattered Intensity Along the Superficial 2mm Depth of the Preparation Walls
Description: Presence of elevated backscattered intensity along the superficial 2mm depth walls of the restoration, which indicates presence of debonding, will be computed as percentage volume of the restoration at every evaluation time point, i.e. baseline, 6 months and 18 months post-operative. Outcome is reported in units of percentage area.
Time Frame: Baseline
Measure: Mean (Standard Error); unit: Percentage
Arm/Group | 90-degree Cavosurface Angle Cavity Margin | Wide-bevel Cavity Margin
Number analyzed (Participants) | 18 | 18
Percentage | 16.20 (4.85) | 7.43 (5.30)

ADVERSE EVENTS:
Time Frame: 18 months
Description: The interventions in both arms are topical one-surface dental resin composite restorations and there are no systemic interventions. Hence the number of participants at risk for All-Cause Mortality and Serious Adverse Events is zero.
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 1/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=18) | Group 2 (N=18)
Discomfort upon biting on the tooth with dental restoration (Surgical and medical procedures) | 1 | 2 — Patient experienced discomfort upon biting on the tooth with the dental restoration about one week after restoration was done. The discomfort was relieved when pressure point was removed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/22/NCT05145322/Prot_SAP_002.pdf
  • Informed Consent Form (2021-12-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT05145322/ICF_001.pdf